CLINICAL TRIAL: NCT06219902
Title: A Randomized, Double-blind, Placebo- and Active-controlled, 4-period, Crossover Study to Investigate Effects of Elinzanetant on Simulated Driving Performance and Cognitive Function in Healthy Women
Brief Title: A Study to Learn if Elinzanetant Affects the Ability to Drive and Brain Function in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 22653
Record Dates: First submitted 2023-12-21; First posted 2024-01-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men; Hot Flashes
Keywords: Driving performance,; Cognitive function
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Hot Flashes | interventions — zopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment sequences A-C-D-B (Experimental): Treatment A (elinzanetant dose A). Treatment B (elinzanetant dose B). Treatment C (zopiclone 7.5 mg). Treatment D (placebo).
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo to elinzanetant; Drug: Zopiclone; Drug: Placebo to zopiclone
- Treatment sequences B-D-C-A (Experimental): Treatment A (elinzanetant dose A). Treatment B (elinzanetant dose B). Treatment C (zopiclone 7.5 mg). Treatment D (placebo).
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo to elinzanetant; Drug: Zopiclone; Drug: Placebo to zopiclone
- Treatment sequences C-B-A-D (Experimental): Treatment A (elinzanetant dose A). Treatment B (elinzanetant dose B). Treatment C (zopiclone 7.5 mg). Treatment D (placebo).
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo to elinzanetant; Drug: Zopiclone; Drug: Placebo to zopiclone
- Treatment sequences D-A-B-C (Experimental): Treatment A (elinzanetant dose A). Treatment B (elinzanetant dose B). Treatment C (zopiclone 7.5 mg). Treatment D (placebo).).
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo to elinzanetant; Drug: Zopiclone; Drug: Placebo to zopiclone

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Oral administration of multiple doses of elinzanetant.
Drug: Placebo to elinzanetant — Oral administration
Drug: Zopiclone — Oral administration
Drug: Placebo to zopiclone — Oral administration

SUMMARY:
Researchers are looking for a better way to treat vasomotor symptoms (VMS), also known as hot flashes.

Hot flashes are intense and sudden feelings of heat along with sweating and reddening of the skin. These are common for women going through the menopause but can also occur in men. Such symptoms are called VMS and are caused by changes in sex hormone levels.

The study treatment, elinzanetant, is being tested for the treatment of VMS in both men and women. It works by blocking the activity of a substance called neurokinin, which is thought to play a role in starting hot flashes.

Elinzanetant may cause lasting effects like sleepiness and tiredness. Such effects may make driving unsafe.

The main purpose of this study is to learn how elinzanetant affects the ability to drive the next day in healthy women.

For this, researchers will study participants' ability to keep a stable position within their lane while driving on a straight road on a computer-based driving test (also known as a driving simulator).

In this study, participants will take 2 different doses of elinzanetant, another drug called zopiclone, and matching placebos to these drugs.

Zopiclone helps treat sleeping problems. A placebo looks like a study drug but does not have any medicine in it.

Participants will take elinzanetant, zopiclone, and their matching placebos by mouth.

This study will have 4 treatment periods with each period lasting 6 days. In each period, participants will receive one of the following treatments in an order assigned to them randomly (by chance):

* dose A of elinzanetant and a zopiclone placebo
* dose B of elinzanetant and a zopiclone placebo
* zopiclone 7.5 milligrams (mg) and elinzanetant placebo
* elinzanetant placebo and zopiclone placebo

Each participant will be in the study for around 15 weeks with up to 6 visits to the study site.

Participants will visit the study site:

* once before the treatment starts, so the study doctors and their team can check on their health and confirm if the participant can join the study
* once in each of the 4 treatment periods for a 6-day stay at the study site with a gap of 14 days between each period. During each stay, they will take the assigned treatment from Days 1 to 5 and the driving test on Days 2 and 6
* once, 2 to 3 days after their last treatment so the study doctors and their team can check on their health

During the study, the doctors and their study team will:

* check participants' health by performing tests such as blood and urine tests, and checking heart health using an electrocardiogram (ECG)
* check the participants' ability to drive and their brain function and level of sleepiness using different tests including a driving simulator test
* check the level of the study drugs in participants' blood
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think they are related to the study treatment or not.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40 to 65 years, inclusive, at signing of informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, blood pressure, pulse rate and electrocardiogram (ECG).
* Participant has a regular sleep pattern, is not engaged in shift-work, and in general, has at least 7 hours of sleep each night (bedtime occurs between 21:00 and 24:00 hours).
* Participant possesses a valid driver's license and is an active driver. Drives a minimum of 8,000 kilometers per year for the previous 3 years.

Exclusion Criteria:

* Relevant diseases within the last 4 weeks prior to the first administration of study intervention, including febrile illness.
* A history within 2 years of, or current treatment for, a sleeping disorder (including excessive snoring, obstructive sleep apnea), or a chronic painful condition that interferes with the participant's sleep.
* Abnormal finding in the physical examination, ECG, blood pressure, pulse rate or clinical laboratory results at Screening, that are considered clinically significant by the investigator.
* Use of any medication of dietary supplement which may affect central nervous system (CNS) function and may confound the pharmacodynamic assessments of the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Simulated driving performance as measured by SDLP using CRCDS-MiniSim | Approximately 9 hours after last dose
  SDLP: standard deviation of lateral position. CRCDS-MiniSim: Cognitive Research Corporation's Driving Simulator-MiniSim.

SECONDARY OUTCOMES:
Lane Exceedance: Number of Exceedance. | Approximately 9 hours after last dose
Lane Exceedance: Maximum Duration of Exceedance. | Approximately 9 hours after last dose
Lane Exceedance: Area of Exceedance. | Approximately 9 hours after last dose
Excessive Speed Count | Approximately 9 hours after last dose
Average Speed and Speed Deviation | Approximately 9 hours after last dose
Driving safety measures: Total number of excessive Ay (cornering speed threshold-exceeded) | Approximately 9 hours after last dose
Driving safety measures: Total number of collisions | Approximately 9 hours after last dose
Divided Attention: Correct responses; Omission Errors; Commission Errors; Reaction Time; Standard Deviation of Reaction Time | Approximately 9 hours after last dose
CogScreen Symbol Digit Coding Test: Number of Correct responses | Approximately 9 hours after last dose
  CogScreen Symbol Digit Coding test is a computer analogue of the conventional digit symbol-substitution task found in the revised Wechsler intelligence scales.
CogScreen Symbol Digit Coding Test: Response Accuracy (percentage of correct responses) | Approximately 9 hours after last dose
CogScreen Symbol Digit Coding Test: Standard Deviation of Reaction Time | Approximately 9 hours after last dose
Karolinska Sleepiness Scale (KSS) Score | Approximately 9 hours after last dose
  The KSS measures an individual's subjective level of sleepiness. Participants indicate their level of alertness versus sleepiness according to a 9-point scale, ranging from "extremely alert" to "extremely sleepy - fighting sleep".
Participant's self-reported Readiness to Drive | Approximately 9 hours after last dose
  Prior to driving, the participant will be asked a simple question as to whether they feel safe to drive ("Right now do you feel safe to drive?"). Participant will answer "yes" or "no".
Self-report of motivation and appraisal of driving performance using VAS | Approximately 9 hours after last dose
  Participants will record their response to each question by drawing a vertical line on a 100-mm horizontal, linear VAS printed on paper.
  For the self-assessment of driving performance, one end of the line is marked "Not Satisfactory" and the other end of the line is marked "Satisfactory".
  For the motivation item, 1 end of the line is marked "Not Motivated" and the other end is marked "Motivated".
  Scores on the 100-mm linear scale will be measured to the nearest millimeter from the left with a ruler.

CONTACTS AND LOCATIONS:
Locations (1):
- AltaSciences, Mount Royal, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Francke K, Klein S, Burke J, Schultze-Mosgau MH, Kay G. The Effects of Elinzanetant on Simulated Driving Performance in Healthy Women: A Randomized Phase I Study. Clin Transl Sci. 2025 Jul;18(7):e70282. doi: 10.1111/cts.70282. PMID 40569207